CLINICAL TRIAL: NCT04522999
Title: An Objective Study to Evaluate the Ability of Photobiomodulation to Improve Electroretinogram Outcomes in Subjects With Dry Age-Related Macular Degeneration
Brief Title: Study of Photobiomodulation Effect on Electroretinogram Outcomes in Dry Age-Related Macular Degeneration
Acronym: ELECTROLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiThera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP007
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Photobiomodulation (Experimental): Valeda™ Light Delivery System
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — The Valeda™ Light Delivery System

SUMMARY:
To evaluate the ability of Photobiomodulation (PBM) treatment using the Valeda® Light Delivery System to improve Electroretinogram (ERG) outcomes in subjects with dry Age-related Macular Degeneration (AMD).

DETAILED DESCRIPTION:
This study is an open label, prospective pilot study to evaluate retinal function after PBM treatment in eyes with dry AMD using ERG. The target enrollment is 15 subjects in up to two sites in the US. All subjects will receive PBM Treatment.

Subjects will receive three PBM treatments per week for three weeks for a total of nine sessions over 3 weeks.

The primary analysis will examine multi-focal ERG function changes from baseline to Month 1. Secondary analyses will examine multi-focal ERG function change from baseline to Month 3 and 6. Other endpoints will include other functions of ERG, ETDRS Visual Acuity, Contrast Sensitivity, Perimetry, Color Vision test and the Amsler grid test.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 50 years of age at Screening visit
* ETDRS BCVA letter score of between 50* and 75* (Snellen equivalent of 20/100 to 20/32)
* Diagnosis of dry AMD
* Able to communicate well with the Investigator and able to understand and comply with the requirements of the study
* Informed of the nature of this study and has provided written, informed consent in accordance with institutional, local and national regulatory guidelines

Exclusion Criteria:

* Current or history of neovascular maculopathy
* Presence of center involving GA within the central ETDRS 1 mm diameter at Screening
* Media opacities, including cataracts, which might interfere with visual acuity or imaging in the study eye(s)
* Posterior capsule opacification, which might interfere with visual acuity or imaging in the study eye(s)
* Invasive eye surgery (e.g. cataract, capsulotomy) on a qualifying eye within three 3 months prior to Screening
* Visually significant disease in any ocular structure apart from dry AMD
* Serious medical illness that will prevent the subject from performing study activities
* Presence of or history of malignancy within the past 5 years
* Presence or history of known light sensitivity to yellow light, red light, or near infrared radiation (NIR), or if they have a history of light activated CNS disorders (e.g. epilepsy, migraine)
* History of neurologic condition known to affect visual function
* History of drug, alcohol or substance abuse within 3 months prior to Screening
* Participation in any other clinical study at time of screening, or has received an investigational drug or treatment with an investigational device within 3 months prior to Screening
* In the opinion of the Investigator, is unlikely to comply with the study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
ERG function | 3 months
  ERG assessments (Multifocal ERG (mfERG), Photopic Negative Response (PhNR), Multi-luminance Flicker ERG (ML-FERG) and Fixed-luminance Flicker ERG (FL-FERG)) will provide an output of retinal function.

OTHER OUTCOMES:
ETDRS Visual Acuity | 3 months
  Measurement of Visual function.
Mars Contrast Sensitivity | 3 months
  Measurement of Visual function.

CONTACTS AND LOCATIONS:
Locations (1):
- Perich Eye Center, New Port Richey, Florida, United States